CLINICAL TRIAL: NCT05099289
Title: Parasternal Access for ShockS and Pacing With an acUtely Placed Less-invasive Lead for EV-ICD (PASS PULL EV-ICD) Study
Acronym: PASS PULL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtaCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DOC-10154
Record Dates: First submitted 2021-09-29; First posted 2021-10-29 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Ventricular Arrhythmia; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: Ventricular Defibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AtaCor EV-ICD Lead System (Experimental): Subjects inserted with the AtaCor EV-ICD Lead Model AC-7000
  Interventions: Device: AtaCor EV-ICD Lead

INTERVENTIONS:
Device: AtaCor EV-ICD Lead — Subjects will receive the AtaCor EV-ICD Lead being evaluated in the study.

SUMMARY:
The PASS PULL EV-ICD Study is a prospective, multi-center, single-arm study without concurrent or historical controls. This initial concept feasibility study is primarily intended to demonstrate that the EV-ICD Lead can be safely positioned within the anterior mediastinum as intended using the AtaCor delivery system. The study will secondarily characterize the ability for the EV-ICD Lead to facilitate VF sensing and defibrillation.

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate that the AtaCor EV-ICD Lead can be safely positioned within the anterior mediastinum as intended using the EV-ICD Dilator and EV-ICD Delivery Tool. The study will secondarily characterize the ability for the EV-ICD Lead to facilitate VF sensing and defibrillation.

Up to 3 Investigational Sites will participate with up to 65 subjects enrolled in the study. Patients undergoing de novo or replacement ICD procedure will be eligible for participation. Study participation requires acute evaluation of the EV-ICD Lead during the index procedure. Echocardiography will be used to evaluate any new or worsening pericardial effusions. A follow-up visit will occur 7-10 days post-removal via phone, video call, or in-person. Participation will end after completion of the 7-10 days post-removal visit. The Study is expected to last up to 3 months for enrollment.

ELIGIBILITY:
Inclusion criteria

1. At least 18 years old
2. Indicated for de novo or replacement ICD procedure

Exclusion criteria

1. NYHA IV functional class
2. BMI ≥ 35 kg/m2
3. Inotropic therapy in past 180 days
4. Subjects with a hemodynamically unstable intrinsic heart rate that requires continual ventricular pacing
5. Presence or planned use of subcutaneous coils/arrays, epicardial patches or epicardial pace/sense leads
6. Subjects on anticoagulation/antiplatelet therapy that cannot be temporarily discontinued for the procedure
7. Logistical or safety related circumstances that may prevent data collection or follow-up
8. Participation in any concurrent clinical study without prior written approval from the Sponsor
9. Inability to give an informed consent to participate in the Study

   Known prior history for any of the following:
10. Structural abnormalities of the heart that may increase risk of the study procedure or an obstructed/restricted pathway into the mediastinum for the EV-ICD Dilator, EV-ICD Delivery Tool and EV-ICD Lead as assessed from available CT or Echocardiography.
11. Uncontrolled paroxysmal, persistent or permanent atrial fibrillation
12. Median or partial sternotomy
13. Surgery with disruption of the lung, pericardium or connective tissue between the sternum and pericardium
14. Significant anatomic derangement of or within the thorax (e.g., pectus excavatum, significant scoliosis)
15. Thoracic radiation therapy, pneumothorax, pneumomediastinum or other medical treatments/conditions which may complicate the EV-ICD Lead insertion procedure
16. Pericardial disease, pericarditis and mediastinitis
17. Medical treatments, surgeries or conditions that increase the potential for pericardial adhesions
18. FEV1 < 1.0 Liter
19. Surgically corrected congenital heart disease (not including catheter-based procedures)
20. Allergies to the device materials as listed in the Instructions for Use (IFU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of SADEs | Up to 10 days post-procedure
  Incidence of Serious Adverse Device Effects (SADEs)
Rate of Insertion Success | Procedure
  Defined as the ability to deploy the lead in a position within the mediastinum that is suitable for defibrillation testing and does not result in one (1) or more SADEs

SECONDARY OUTCOMES:
Functionality - Lowest Defibrillation Conversion Energy | Procedure
  Lowest Defibrillation Conversion Energy (J)
Observational: Incidence of ADEs | Up to 10 days post-procedure
  Incidence of Adverse Device Effects (ADEs), Overall and Individual

CONTACTS AND LOCATIONS:
Overall Officials: Martin C Burke, DO, Principal Investigator — AtaCor Medical, Inc.
Locations (1):
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No